CLINICAL TRIAL: NCT04075825
Title: A Follow-up of a Phase 3 Study to Evaluate the Long-term Safety and Efficacy of Darvadstrocel in the Treatment of Complex Perianal Fistula in Subjects With Crohn's Disease Who Have Participated in ADMIRE II Study
Brief Title: Long-term Follow-up Study With Darvadstrocel in the Treatment of Complex Perianal Fistula
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Darvadstrocel-3003; 2019-000333-39 (EudraCT Number)
Record Dates: First submitted 2019-08-22; First posted 2019-09-03 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Crohn's Disease; Complex Perianal Fistula
Keywords: Drug therapy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants who received darvadstrocel placebo-matching expanded adipose-derived stem cells (eASCs) intralesional injection previously in the ADMIRE-CD II study were observed for efficacy and safety. No drug was administered in this study.
  Interventions: Other: Placebo
- Darvadstrocel (Experimental): Participants who received a single dose of darvadstrocel, 120 million cells, intralesionally previously in the ADMIRE-CD II study were observed for efficacy and safety. No drug was administered in this study.
  Interventions: Biological: Darvadstrocel

INTERVENTIONS:
Other: Placebo — Darvadstrocel placebo-matching eASCs intralesional injection received in previous ADMIRE-CD II study. No drug administration in this study.
  Arms: Placebo
Biological: Darvadstrocel — Allogenic expanded adipose-derived stem cells (eASCs) 5 million cells/ml - suspension for injection darvadstrocel received in previous ADMIRE-CD II study. No drug administration in this study.
  Other Names: Cx601
  Arms: Darvadstrocel

SUMMARY:
The main aim is to follow-up on long term side effect and symptom improvement of Darvadstrocel in the treatment of complex perianal fistula in adults. Participants will not receive any drug in this study.

DETAILED DESCRIPTION:
The drug being tested in this study is called darvadstrocel (Cx601). Darvadstrocel is being tested to treat people who have complex perianal fistula in CD. This study will look at the long-term safety and efficacy of darvadstrocel in the treatment of complex perianal fistula in CD.

The study will enroll approximately 150 patients. Participants who received darvadstrocel or placebo in study ADMIRE-CD II (Cx601-0303, NCT03279081) and who have completed the 52 weeks of the study will be enrolled in this long-term extension study.

This multi-center study will be conducted worldwide. The overall time to participate in this study is 104 weeks (in addition to the 52 weeks on ADMIRE-CD II study). Participants will make multiple visits to the clinic and will be contacted by telephone every 3 months for a follow-up assessment. After unblinding of the ADMIRE-CD II study, the LTE study will be conducted as an open-label study. Participants will remain in the treatment group assigned in the ADMIRE-CD II study.

ELIGIBILITY:
Inclusion Criteria:

1. Has participated in and completed the ADMIRE-CD II (NCT03279081) study (i.e., did not discontinue).

Exclusion Criteria:

1. Has been more than 3 months since the participant completed the ADMIRE-CD II study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (58):
- United States (22):
  - University of California San Francisco, San Francisco, California
  - Cedar-Sinai Medical Center, West Hollywood, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Cleveland Clinic Florida, Fort Lauderdale, Florida
  - University of Miami Hospital, Miami, Florida
  - USF Health South Tampa Center for Advanced Healthcare, Tampa, Florida
  - AdventHealth Tampa, Tampa, Florida
  - Indiana University - Colon and Rectal, Indianapolis, Indiana
  - University of Kansas Medical Center (KUMC) - University of Kansas Liver Center - Hepatology Clinic, Kansas City, Kansas
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Massachussetts General Hospital - Gastroenterology, Boston, Massachusetts
  - Mayo Clinic College of Medicine - Division of Colon and Rectal Surgery - Division of Colon and Rectal Surgery, Rochester, Minnesota
  - Dartmouth Hitchcock Medical Center - Cancer Center, Lebanon, New Hampshire
  - Morristown Medical Center - Gastroenterology, Morristown, New Jersey
  - Northwell Health, Manhasset, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Penn State Hershey Medical Center - Surgery, Hershey, Pennsylvania
  - Brown Surgical Associates,Inc., Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia
  - Virginia Mason Medical Center - Gastroenterology, Seattle, Washington
- Belgium (3):
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams Brabant
  - GZA Sint-Vincentius, Antwerp
- Czechia (2):
  - NH Hospital a.s., Hořovice
  - FN Hradec Kralove, Hradec Králové
- France (7):
  - CHRU de Brabois Hopitaux de Brabois, Vandœuvre-lès-Nancy, Nancy
  - CHRU de Lille - Hopital Claude Huriez - Gastroenterologie, Lille, Nord
  - CHU de Clermont-Ferrand - Estaing, Clermont-Ferrand
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHRU Hopital de Pontchaillou - Maladies De L'Appareil Digesti, Rennes
  - Paris St. Joseph Hospital, Paris, Île-de-France Region
- Hungary (4):
  - Szegedi Tudomanyegyetem Altalanos Orvostudomanyi Kar, Szeged, Csongrád megye
  - MH Egeszsegugyi Kozpont, Budapest, Pest County
  - Semmelweis Egyetem Altalanos Orvostudomanyi Kar, Budapest
  - Debreceni Egyetem Klinikai Kozpont Nagyerdei Campus Gyermekgyogyaszati Klinika, Debrecen
- Israel (4):
  - Rabin Medical Center, Beilinson Hospital -Gastroenterology, Petah Tikva, Central District
  - Hadassah Medical Organization, Hadassah Medical Center, Ein-, Jerusalem, Jerusalem
  - Rambam Medical Centre, Haifa
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (3):
  - AOU Policlinico di Modena - Gastroenterologia, Modena
  - Complesso Integrato Columbus, Universita Cattolica del Sacro Cuore, Roma
  - PU A. Gemelli, Universita Cattolica del Sacro Cuore, Roma
- Poland (2):
  - Centrum Medyczne Melita Medical, Wroclaw, Lower Silesian Voivodeship
  - Wielospecjalistyczny Szpital Medicover, Warsaw
- Spain (11):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - H.U. G.Trias i Pujol, Badalona, Barcelona
  - Parc Tauli Hospital Universitari, Sabadell, Barcelona
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Del Mar, Barcelona
  - Hospital Clinic De Barcelona, Barcelona
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - C.H.U. de Pontevedra, Pontevedra
  - H.U.V. del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b603c4db2bf003ab4a350?idFilter=%5B%22Darvadstrocel-3003%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites globally from 05 November 2019 to 02 April 2024.
Pre-assignment Details: Participants diagnosed with Complex Perianal Fistula in Crohn's Disease (CD) who completed the Week 52 visit in the parent study ADMIRE-CD II (Cx601-0303, NCT03279081) were enrolled. Participants remained in the treatment group (placebo or darvadstrocel) to which they were assigned in ADMIRE-CD II study.
Period: Overall Study
Arm/Group | Placebo | Darvadstrocel
Started | 74 | 76
Completed | 57 | 63
Not Completed | 17 | 13
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Physician Decision | 3 | 1
Not completed — Lost to Follow-up | 5 | 1
Not completed — Participation in New Clinical Trial | 1 | 1
Not completed — Reason Not Specified | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants enrolled in the long-term extension (LTE) study, according to the actual treatment they received in the ADMIRE-CD II study.
  Week 52 of ADMIRE-CD II is the Baseline (Week 0) for this study.
Groups:
- Placebo: Participants who received darvadstrocel placebo-matching eASCs intralesional injection previously in the ADMIRE-CD II study were observed for efficacy and safety. No drug was administered in this study.
- Total: Total of all reporting groups
Arm/Group | Placebo | Darvadstrocel | Total
Number analyzed (Participants) | 74 | 76 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (11.33) | 40.6 (12.04) | 39.8 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 35 | 63
  Male | 46 | 41 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 65 | 62 | 127
  Unknown or Not Reported | 4 | 10 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 73 | 68 | 141
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 7 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered an investigational medicinal product; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a study intervention or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the study intervention or medicinal product.
Time Frame: Baseline (Week 0) up to Week 104 of this study (Week 52 up to Week 156 in relation to ADMIRE-CD II)
Population: Safety Analysis Set included all participants enrolled in the LTE study, according to the actual treatment they received in the ADMIRE-CD II study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darvadstrocel
Number analyzed (Participants) | 74 | 76
Participants | 40 | 43

2. Primary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (TESAEs)
Description: TEAE is defined as: any adverse event emerging/manifesting at or after the initiation of treatment with a study intervention/medicinal product or any existing event that worsens in either intensity/frequency following exposure to the study intervention/medicinal product. Serious adverse event (SAE) is an untoward medical occurrence, significant hazard, contraindication, side effect/precaution that at any dose: results in death, is life-threatening, required in-patient hospitalization/prolongation of existing hospitalization, results in persistent/significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: Baseline (Week 0) up to Week 104 of this study (Week 52 up to Week 156 in relation to ADMIRE-CD II)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darvadstrocel
Number analyzed (Participants) | 74 | 76
Participants | 14 | 11

3. Primary Outcome: Number of Participants With Specific Adverse Events of Special Interest (AESIs)
Description: AESIs are AEs that are not solicited local or systemic AEs, they are predefined AEs that require close monitoring and prompt reporting to the sponsor. Protocol pre-specified AESIs included immunogenicity/allo-immunoreactions, tumorigenicity, ectopic tissue formation and fistula/abscess. In addition, ad hoc AESIs of anaphylactic reaction, hypersensitivity, and malignancy.
Time Frame: Baseline (Week 0) up to Week 104 of this study (Week 52 up to Week 156 in relation to ADMIRE-CD II)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Darvadstrocel
Number analyzed (Participants) | 74 | 76
Participants
  Immunogenicity/Allo-immunoreactions | 3 | 7
  Tumorgenicity | 1 | 3
  Fistula, Abscess | 6 | 7
  Ectopic Tissue Formation | 1 | 0
  Hypersensitivity | 3 | 3
  Anaphylactic Reaction | 0 | 0
  Malignancy | 1 | 2

4. Secondary Outcome: Percentage of Participants Who Achieve Clinical Remission at Weeks 104 and 156 (After IMP Administration in ADMIRE-CD II Study)
Description: Clinical remission is defined as closure of all treated external fistula openings that were draining at baseline of ADMIRE-CD II despite gentle finger compression. Percentages were rounded off to the nearest second decimal place.
Time Frame: At Weeks 52 and 104 of this study (Weeks 104 and 156 in relation to ADMIRE-CD II, respectively)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Darvadstrocel
Number analyzed (Participants) | 74 | 76
percentage of participants
  Week 52 | 36.49 [25.52 to 47.45] | 50.00 [38.76 to 61.24]
  Week 104 | 31.08 [20.54 to 41.63] | 43.42 [32.28 to 54.56]

5. Secondary Outcome: Percentage of Participants Who Achieve Clinical Response at Weeks 104 and 156 (After IMP Administration in ADMIRE-CD II Study)
Description: Clinical response is defined as closure of at least 50% of all treated external fistula openings that were draining at baseline of ADMIRE-CD II despite gentle finger compression. Percentages were rounded off to the nearest second decimal place.
Time Frame: At Weeks 52 and 104 of this study (Weeks 104 and 156 in relation to ADMIRE-CD II, respectively)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Darvadstrocel
Number analyzed (Participants) | 74 | 76
percentage of participants
  Week 52 | 40.54 [29.35 to 51.73] | 56.58 [45.44 to 67.72]
  Week 104 | 32.43 [21.77 to 43.10] | 47.37 [36.14 to 58.59]

6. Secondary Outcome: Percentage of Participants With Relapse at Week 156 After Achieving Combined Remission at Week 52 of ADMIRE-CD II
Description: Relapse is defined as participants who were in combined remission at Week 52 of ADMIRE-CD II and who have either reopening of any of the treated fistula(s) external openings with active drainage as clinically assessed or, the development of a perianal fluid collection >2 cm of the treated perianal fistulas confirmed by centrally read magnetic resonance imaging (MRI) assessment. Combined remission at Week 52 was defined as clinically assessed closure of all treated external openings that were draining at baseline of ADMIRE-CD II, despite gentle finger compression, and absence of collection(s) >2 cm (in at least 2 dimensions) of the treated perianal fistula(s) confirmed by blinded central MRI assessment. Percentages were rounded off to the nearest second decimal place.
Time Frame: At Week 104 of this study (Week 156 in relation to ADMIRE-CD II)
Population: Safety Analysis Set included all participants enrolled in the LTE study, according to the actual treatment they received in the ADMIRE-CD II study. . Overall number analyzed is the number of participants who were in combined remission at Week 52 of ADMIRE-CD II.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Darvadstrocel
Number analyzed (Participants) | 42 | 40
percentage of participants | 54.76 [39.71 to 69.81] | 42.50 [27.18 to 57.82]

7. Secondary Outcome: Percentage of Participants Who Achieve Combined Remission at Week 156 (After IMP Administration in ADMIRE-CD II Study)
Description: Combined remission of complex perianal fistula(s) is defined as the clinical assessment of closure of all treated external openings that were draining at baseline of ADMIRE-CD II, despite gentle finger compression, and absence of collection(s) >2 cm (in at least 2 dimensions) of the treated perianal fistula(s) confirmed by centrally read blinded MRI assessment. Percentages were rounded off to the nearest second decimal place.
Time Frame: At Week 104 of this study (Week 156 in relation to ADMIRE-CD II)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Darvadstrocel
Number analyzed (Participants) | 74 | 76
percentage of participants | 29.73 [19.32 to 40.14] | 36.84 [26.00 to 47.69]

8. Secondary Outcome: Percentage of Participants With New Anal Abscess in Treated Fistula at Week 156
Description: Percentages were rounded off to the nearest second decimal place.
Time Frame: At Week 104 of this study (Week 156 in relation to ADMIRE-CD II)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Darvadstrocel
Number analyzed (Participants) | 74 | 76
percentage of participants | 9.62 [3.20 to 21.03] | 7.02 [1.95 to 17.00]

9. Secondary Outcome: Change From Baseline of ADMIRE-CD II in Scores of Discharge Items of Perianal Disease Activity Index (PDAI) Score at Weeks 104 and 156
Description: The PDAI is a scoring system to evaluate the severity of perianal CD. From the 5-item instrument, only 'discharge' was used for this outcome measure. Each category is graded on a 5-point Likert scale ranging from no symptoms (score of 0) to severe symptoms (score of 4); a higher score indicates more severe disease.
Time Frame: From Baseline of ADMIRE-CD II up to Weeks 52 and 104 of this study (From Baseline up to Weeks 104 and 156 in relation to ADMIRE-CD II, respectively)
Population: Safety Analysis Set included all participants enrolled in the LTE study, according to the actual treatment they received in the ADMIRE-CD II study. Overall number analyzed is the number of participants with data available at ADMIRE-CD II Baseline. Number analyzed is the number of participants with data available for analyses at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Darvadstrocel
Number analyzed (Participants) | 59 | 67
score on a scale
  ADMIRE-CD II Baseline Score | 1.53 (1.072) | 1.25 (0.893)
  Change from ADMIRE-CD II Baseline up to Week 52 of this study: number analyzed (Participants) | 51 | 61
  Change from ADMIRE-CD II Baseline up to Week 52 of this study | -0.67 (1.178) | -0.56 (1.218)
  Change from ADMIRE-CD II Baseline up to Week 104 of this study: number analyzed (Participants) | 45 | 56
  Change from ADMIRE-CD II Baseline up to Week 104 of this study | -0.67 (1.279) | -0.50 (1.128)

10. Secondary Outcome: Change From Baseline of ADMIRE-CD II in Scores of Pain Items of Perianal Disease Activity Index (PDAI) Score at Weeks 104 and 156
Description: The PDAI is a scoring system to evaluate the severity of perianal CD. From the 5-item instrument, only 'pain' was used for this outcome measure. Each category is graded on a 5-point Likert scale ranging from no symptoms (score of 0) to severe symptoms (score of 4); a higher score indicates more severe disease.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Darvadstrocel
Number analyzed (Participants) | 59 | 67
score on a scale
  ADMIRE-CD II Baseline Score | 1.25 (1.060) | 1.06 (0.936)
  Change from ADMIRE-CD II Baseline up to Week 52 of this study: number analyzed (Participants) | 51 | 61
  Change from ADMIRE-CD II Baseline up to Week 52 of this study | -0.49 (1.391) | -0.54 (1.010)
  Change from ADMIRE-CD II Baseline up to Week 104 of this study: number analyzed (Participants) | 45 | 56
  Change from ADMIRE-CD II Baseline up to Week 104 of this study | -0.56 (1.271) | -0.45 (1.060)

ADVERSE EVENTS:
Time Frame: Up to 104 weeks in this study (From Week 52 to Week 156 in relation to ADMIRE-CD II)
Description: Safety Analysis Set included all participants enrolled in the LTE study, according to the actual treatment they received in the ADMIRE-CD II study.
Arm/Group | Placebo | Darvadstrocel
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/76
Serious Adverse Events (participants affected / at risk) | 14/74 | 11/76
Other Adverse Events (participants affected / at risk) | 11/74 | 14/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=74) | Darvadstrocel (N=76)
Abdominal abscess (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 2 | 3
Anal fistula (Gastrointestinal disorders) | 2 | 1
Anorectal disorder (Gastrointestinal disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 2
Calculus urinary (Renal and urinary disorders) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Fistula discharge (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Terminal ileitis (Gastrointestinal disorders) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=74) | Darvadstrocel (N=76)
COVID-19 (Infections and infestations) | 8 | 9
SARS-CoV-2 test positive (Investigations) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT04075825/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/25/NCT04075825/SAP_001.pdf